CLINICAL TRIAL: NCT05919836
Title: Different Laparoscopic Techniques for Management of Congenital Inguinal Hernia in Pediatrics
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Mario Ayoub Youssef Sorial, Investigator, Assiut University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: lap hernia in pediatrics
Record Dates: First submitted 2023-04-20; First posted 2023-06-26 (Actual); Last update posted 2023-06-26 (Actual); Status verified 2023-06

CONDITIONS: Congenital Inguinal Hernia

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Percutaneous assisted laparoscopic hernia (Active Comparator)
  Interventions: Procedure: Laparoscopic assisted hernia
- Laparoscopic Purse string closure of hernial sac (Active Comparator)
  Interventions: Procedure: Laparoscopic hernia by purse string closure
- Laparoscopic Total dissection of hernial sac (Active Comparator)
  Interventions: Procedure: Total laparoscopic dissection of hernial sac

INTERVENTIONS:
Procedure: Laparoscopic assisted hernia — Percutaneous assisted laparoscopic hernia
  Arms: Percutaneous assisted laparoscopic hernia
Procedure: Laparoscopic hernia by purse string closure — Laparoscopic purse string closure of hernial sac
  Arms: Laparoscopic Purse string closure of hernial sac
Procedure: Total laparoscopic dissection of hernial sac — Total laparoscopic dissection of hernial sac
  Arms: Laparoscopic Total dissection of hernial sac

SUMMARY:
Comparison between multiple approaches of laparoscopic hernia ( percutaneous assisted laparoscopic hernia, purse string closure of hernial sac, total dissection of hernial sac).

DETAILED DESCRIPTION:
In pediatric age, indirect inguinal hernia represents more than 95% of the hernial disease. It is a congenital type, in contrast with adulthood in which acquired forms are more frequently found.

Inguinal hernia repair is one of the most frequently performed surgical procedure in infants and young children. Laparoscopic hernia repair in infancy and childhood is still debatable. There are many techniques available for laparoscopic hernia repair in pediatrics.

Laparoscopic hernial repair is increasingly adopted even for neonates and has achieved a high success rate with low recurrence rate with long-term follow-up. The main advantages of laparoscopy are no incision of the fascia, exploration of the other side in case of bilateral hernia, and visualization and safeguarding of the vas deferens and the spermatic vessels. Moreover, it is advantageous over open technique in case of recurrent hernia. Different modalities of techniques have been used for repair such as needlescopic disconnection of hernia sac, flip flap technique, muscular arch repair, and ring closure.

ELIGIBILITY:
Inclusion Criteria:

* patients in the age limit with congenital inguinal hernia

Exclusion Criteria:

* recurrent hernias
* cases inwhich laparoscopic surgery is contraindicated
* cases with collagen defect diseases

Ages: 1 Month to 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 69 (Estimated)
Dates: Start 2023-09 (Estimated); Primary Completion 2025-04 (Estimated); Study Completion 2025-06 (Estimated)

PRIMARY OUTCOMES:
Operative time | 4 months
  Comparison between operative time in the three approaches
Early recurrence | 4 months
  Comparison between early recurrence of hernia in the three approaches
Post operative pain duration | 4 months
  Comparison between post operative pain duration between the three approaches

IPD SHARING:
Plan to Share IPD: Undecided